CLINICAL TRIAL: NCT00532259
Title: Phase II Safety and Efficacy Study of the Monoclonal Antibody CT-011 in Patients With Diffuse Large B-Cell Lymphoma Following Autologous Stem Cell Transplantation
Brief Title: CT-011 MAb in DLBCL Patients Following ASCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CureTech Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-2007-01
Record Dates: First submitted 2007-09-19; First posted 2007-09-20 (Estimated); Results first posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Lymphoma, Large Cell, Diffuse; Lymphoma, Mixed Cell, Diffuse; Primary Mediastinal Large B-Cell Lymphoma
Keywords: Lymphoma, Large B-Cell, Diffuse; Transformed Follicular Lymphoma; Stem cell transplantation; Relapsed; Refractory
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Recurrence | interventions — pidilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CT-011 (Experimental): The monoclonal antibody termed CT-011 (currently, pidilizumab).
  Interventions: Drug: CT-011

INTERVENTIONS:
Drug: CT-011 — IV infusion of 1.5 mg/kg of CT-011 on Day 1(60 to 90 days post autologous PBSCT). Treatment was repeated every 42 days for a total of three courses with treatment visits on Days 1, 43, and 85.
  Other Names: Pidilizumab

SUMMARY:
Autologous peripheral blood stem cell transplantation combined with high dose chemotherapy is the treatment of choice given to patients with diffuse large-B cell lymphoma (DLBCL) following relapse of the disease. Although many people are cured of their lymphoma with this therapy, the disease comes back in a certain proportion of patients. The purpose of this study is to test the safety and effectiveness of the monoclonal antibody, CT-011, in patients with DLBCL who have received autologous peripheral blood stem cell transplantation. All final eligible patients will receive an IV infusion of CT-011 on Day 1 (30 to 90 days post autologous PBSCT). Treatment will be repeated every 42 days for a total of three courses with treatment visits on Days 1, 43, and 85. Follow-up for safety and clinical outcome will be conducted throughout the study till 18 months post autologous PBSCT. Approximately 70 patients will participate in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's age is 18 years or older, both genders.
2. Confirmed Diffuse Large B-cell Lymphoma, transformed follicular lymphoma, diffuse mixed cell lymphoma or primary mediastinal large cell lymphoma with B-cell lineage.
3. The lymphoma is chemosensitive.
4. The lymphoma did not progress since pre-transplant chemotherapy.
5. ECOG performance status 0-1.

Exclusion Criteria:

1. Serious other illness.
2. Active autoimmune disease.
3. Type 1 diabetes.
4. Known immune deficiency.
5. Clinical evidence of primary or secondary brain or spinal cord involvement by lymphoma.
6. Active bacterial, fungal, or viral infection.
7. Positive HIV, Hepatitis B surface antigen plus viremia, or Hepatitis C antibody plus viremia.
8. Pregnant or nursing (positive pregnancy test).
9. Other concurrent clinical study or investigational therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2007-10; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leo I Gordon, MD, Principal Investigator — Northwestern University Feinberg School of Medicine; Arnon Nagler, MD, Principal Investigator — Chaim Sheba Medical Center
Locations (27):
- United States (20):
  - Moores UCSD Cancer Center, La Jolla, California
  - Scripps Cancer Center, San Diego, California
  - Emory University-Winship Cancer Institute, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northwestestern Memorial Hospital, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Karmanos Cancer Institute, Detroit, Michigan
  - University of North Carolina, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Ohio State University, Colombus, Ohio
  - Temple University, Philadelphia, Pennsylvania
  - The University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Cancer Center of the Carolinas, Greenville, South Carolina
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Baylor Sammons Cancer Center, Dallas, Texas
  - M.D. Anderson Cancer Center, Houston, Texas
- India (4):
  - Jaslok Hospital and Research Centre, Mumbai, Maharashtra
  - Deenanath Mangeshkar Hospital and Research Centre, Pune, Maharashtra
  - Gujarat Cancer and Research Institute, Ahmedabad
  - Rajiv Gandhi Cancer Institute and Research Centre, Delhi
- Israel (3):
  - Rambam Medical Center, Haifa
  - Hadassah Medical Organization, Jerusalem
  - Chaim Sheba Medical Center, Tel Hashomaer, Ramat Gan

REFERENCES:
- [Derived] Armand P, Nagler A, Weller EA, Devine SM, Avigan DE, Chen YB, Kaminski MS, Holland HK, Winter JN, Mason JR, Fay JW, Rizzieri DA, Hosing CM, Ball ED, Uberti JP, Lazarus HM, Mapara MY, Gregory SA, Timmerman JM, Andorsky D, Or R, Waller EK, Rotem-Yehudar R, Gordon LI. Disabling immune tolerance by programmed death-1 blockade with pidilizumab after autologous hematopoietic stem-cell transplantation for diffuse large B-cell lymphoma: results of an international phase II trial. J Clin Oncol. 2013 Nov 20;31(33):4199-206. doi: 10.1200/JCO.2012.48.3685. Epub 2013 Oct 14. PMID 24127452

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 22 February 2008 (first patient enrolled) to 02 June 2011 (last patient completed) The study was carried out in medical centers
Groups:
- CT-011 Antibody: CT-011 : IV infusion of 1.5 mg/kg of CT-011 on Day 1(30 to 90 days post autologous PBSCT). Treatment was repeated every 42 days for a total of three courses with treatment visits on Days 1, 43, and 85.
Period: Overall Study
Arm/Group | CT-011 Antibody
Started | 72
Completed | 40
Not Completed | 32
Not completed — Withdrawal by Subject | 2
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Lack of Efficacy | 21
Not completed — Lost to Follow-up | 3
Not completed — Physician Decision | 3
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | CT-011 Antibody
Number analyzed (Participants) | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 57
  >=65 years | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 48
Region of Enrollment [Number; unit: participants]
  United States | 58
  Israel | 10
  India | 3
  Chile | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: PFS (progression-free survival ) will be determined at the eligible patient populations
Time Frame: 16 months following the first CT-011 administration (approximately 18 months following autologous PBSCT).
Population: Patients who did not meet key study entry criteria were excluded from the eligible data set.
Measure: Number (90% Confidence Interval); unit: Percent
Arm/Group | CT-011 Antibody
Number analyzed (Participants) | 66
Percent | 72 [60 to 82]

2. Secondary Outcome: Overall Survival
Time Frame: within 16 months following the first CT-011 treatment (18 months following autologous PBSCT).
Measure: Number (90% Confidence Interval); unit: Percent
Arm/Group | CT-011
Number analyzed (Participants) | 66
Percent | 85 [78 to 93]

ADVERSE EVENTS:
Time Frame: 3 years, 3 months
Arm/Group | CT-011 Antibody
Serious Adverse Events (participants affected / at risk) | 23/72
Other Adverse Events (participants affected / at risk) | 69/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CT-011 Antibody (N=72)
Neutropenia (Blood and lymphatic system disorders) | 6 (7)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (4)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Herpes zoster disseminated (Infections and infestations) | 1 (1)
H1n1 Influenza (Infections and infestations) | 1 (1)
Lobar pneumonia (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Vascular injury (Injury, poisoning and procedural complications) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 1 (1)
Pelvic Fracture (Injury, poisoning and procedural complications) | 1 (1)
Head Injury (Injury, poisoning and procedural complications) | 1 (1)
Biopsy Lymph Gland (Investigations) | 1 (1)
Laparoscopy (Investigations) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 1 (1)
Abdominal Hernia Repair (Surgical and medical procedures) | 1 (1)
Knee Arthroplasty (Surgical and medical procedures) | 1 (1)
Small Intestinal Resection (Surgical and medical procedures) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.4% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | CT-011 Antibody (N=72)
Anaemia (Blood and lymphatic system disorders) | 5/69 (6)
Leukopenia (Blood and lymphatic system disorders) | 5 (7)
Lymphopenia (Blood and lymphatic system disorders) | 5 (5)
Lymphadenopathy (Blood and lymphatic system disorders) | 3 (3)
Neutropenia (Blood and lymphatic system disorders) | 13 (18)
Idiopathic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (11)
Palpitations (Cardiac disorders) | 1 (1)
Mitral Valve Incompetence (Cardiac disorders) | 1 (1)
Left Ventricular Dysfunction (Cardiac disorders) | 1 (1)
Sinus Bradycardia (Cardiac disorders) | 1 (1)
Sinus Tachycardia (Cardiac disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 3 (3)
Blindness (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Conjunctivitis Allergic (Eye disorders) | 1 (1)
Eye Oedema (Eye disorders) | 1 (1)
Periorbital Oedema (Eye disorders) | 2 (2)
Eye Pruritus (Eye disorders) | 1 (1)
Vision Blurred (Eye disorders) | 1 (1)
Visual Impairment (Eye disorders) | 1 (1)
Rectal Ulcer (Gastrointestinal disorders) | 1 (1)
Hiatus Hernia (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 12 (19)
Duodenal Ulcer (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Flatulence (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 4 (4)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 (2)
Abdominal Discomfort (Gastrointestinal disorders) | 2 (2)
Defaecation Urgency (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 8 (9)
Vomiting (Gastrointestinal disorders) | 4 (6)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 2 (3)
Mouth Haemorrhage (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Fatigue (General disorders) | 18 (21)
Pyrexia (General disorders) | 8 (10)
Chills (General disorders) | 2 (2)
Feeling Cold (General disorders) | 1 (1)
General Physical Health Deterioration (General disorders) | 1 (1)
Influenza Like Illness (General disorders) | 1 (1)
Local Swelling (General disorders) | 1 (1)
Oedema Peripheral (General disorders) | 1 (1)
Chest Discomfort (General disorders) | 1 (1)
Chest Pain (General disorders) | 1 (2)
Facial Pain (General disorders) | 2 (2)
Pain (General disorders) | 3 (3)
Cholelithiasis (Hepatobiliary disorders) | 2 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1)
Hepatitis (Hepatobiliary disorders) | 1 (1)
Seasonal Allergy (Immune system disorders) | 1 (1)
Hypogammaglobulinaemia (Immune system disorders) | 1 (1)
Enterocolitis Infectious (Infections and infestations) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1)
Candidiasis (Infections and infestations) | 1 (1)
Clostridial Infection (Infections and infestations) | 1 (1)
Tooth Abscess (Infections and infestations) | 1 (1)
Ear Infection (Infections and infestations) | 1 (2)
Fungal Infection (Infections and infestations) | 1 (1)
Gastrointestinal Fungal Infection (Infections and infestations) | 1 (1)
Oral Fungal Infection (Infections and infestations) | 1 (1)
Helicobacter Infection (Infections and infestations) | 1 (1)
Herpes Zoster (Infections and infestations) | 4 (4)
Oral Herpes (Infections and infestations) | 1 (1)
Abscess Limb (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 3 (3)
Bronchitis (Infections and infestations) | 4 (4)
Lung Infection (Infections and infestations) | 1 (2)
Pneumonia (Infections and infestations) | 1 (1)
Skin Infection (Infections and infestations) | 1 (1)
Chronic Sinusitis (Infections and infestations) | 1 (2)
Nasopharyngitis (Infections and infestations) | 2 (3)
Rhinitis (Infections and infestations) | 2 (2)
Sinusitis (Infections and infestations) | 6 (9)
Upper Respiratory Tract Infection (Infections and infestations) | 14 (15)
Urinary Tract Infection (Infections and infestations) | 3 (3)
Viral Rash (Infections and infestations) | 1 (1)
Procedural Nausea (Injury, poisoning and procedural complications) | 1 (1)
Foot Fracture (Injury, poisoning and procedural complications) | 1 (1)
Muscle Strain (Injury, poisoning and procedural complications) | 1 (1)
Anxiety Postoperative (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Procedural Hypotension (Injury, poisoning and procedural complications) | 1 (1)
Procedural Pain (Injury, poisoning and procedural complications) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 1 (1)
Blood Cholesterol Increased (Investigations) | 1 (2)
Activated Partial Thromboplastin Time Prolonged (Investigations) | 4 (7)
International Normalised Ratio (Investigations) | 1 (1)
International Normalised Ratio Increased (Investigations) | 1 (1)
Electrocardiogram Abnormal (Investigations) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 3 (3)
Hepatic Enzyme Increased (Investigations) | 1 (1)
Liver Function Test Abnormal (Investigations) | 1 (1)
Blood Phosphorus Decreased (Investigations) | 1 (1)
Blood Potassium Decreased (Investigations) | 1 (1)
Blood Sodium Decreased (Investigations) | 1 (1)
Blood Sodium Increased (Investigations) | 1 (1)
Serum Ferritin Increased (Investigations) | 1 (1)
Lymph Node Palpable (Investigations) | 1 (1)
Weight Decreased (Investigations) | 2 (2)
Weight Increased (Investigations) | 3 (3)
Blood Thyroid Stimulating Hormone Increased (Investigations) | 1 (1)
Platelet Count Decreased (Investigations) | 5 (5)
Haemoglobin Decreased (Investigations) | 9 (9)
Blood Creatinine Increased (Investigations) | 2 (2)
Blood Testosterone Decreased (Investigations) | 1 (1)
Biopsy Prostate Normal (Investigations) | 1 (1)
Blood Alkaline Phosphatase Increased (Investigations) | 2 (3)
Neutrophil Count Decreased (Investigations) | 6 (7)
White Blood Cell Count Decreased (Investigations) | 9 (12)
White Blood Cell Count Increased (Investigations) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 5 (5)
Hypocalcaemia (Metabolism and nutrition disorders) | 2 (2)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 4 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 9 (12)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatraemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Bursa Disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (5)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3 (4)
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Diffuse Large B-Cell Lymphoma Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Haemorrhage Intracranial (Nervous system disorders) | 1 (1)
Subarachnoid Haemorrhage (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 3 (6)
Syncope (Nervous system disorders) | 1 (1)
Viith Nerve Paralysis (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 6 (8)
Sinus Headache (Nervous system disorders) | 1 (1)
Memory Impairment (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 6 (6)
Presyncope (Nervous system disorders) | 2 (2)
Muscle Contractions Involuntary (Nervous system disorders) | 2 (2)
Paraesthesia (Nervous system disorders) | 2 (2)
Neuropathy Peripheral (Nervous system disorders) | 5 (5)
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Restless Legs Syndrome (Nervous system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 7 (7)
Libido Decreased (Psychiatric disorders) | 2 (2)
Dysuria (Renal and urinary disorders) | 2 (2)
Micturition Urgency (Renal and urinary disorders) | 1 (1)
Renal Failure (Renal and urinary disorders) | 3 (3)
Renal Cyst (Renal and urinary disorders) | 1 (1)
Glycosuria (Renal and urinary disorders) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1)
Nipple Pain (Reproductive system and breast disorders) | 1 (1)
Erectile Dysfunction (Reproductive system and breast disorders) | 1 (1)
Sexual Dysfunction (Reproductive system and breast disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 12 (14)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Allergic Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus Congestion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Night Sweats (Skin and subcutaneous tissue disorders) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Hypoaesthesia Facial (Skin and subcutaneous tissue disorders) | 1 (1)
Macule (Skin and subcutaneous tissue disorders) | 1 (1)
Pain Of Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Scar Pain (Skin and subcutaneous tissue disorders) | 1 (1)
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2)
Rash Erythematous (Skin and subcutaneous tissue disorders) | 3 (3)
Nail Discolouration (Skin and subcutaneous tissue disorders) | 1 (1)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (4)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 6 (7)
Rash Macular (Skin and subcutaneous tissue disorders) | 2 (2)
Lymphadenectomy (Surgical and medical procedures) | 1 (1)
Aortic Aneurysm (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hot Flush (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 3 (3)
Hypotension (Vascular disorders) | 7 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No